CLINICAL TRIAL: NCT05408871
Title: Pilot Study of Non-invasive Measurement of PD-L1 Levels With Positron Emission Tomography (PET) in Head and Neck Malignancies and Intracranial Metastases
Brief Title: Non-invasive Measurement of PD-L1 Levels With Positron Emission Tomography (PET) in Head and Neck Malignancies and Intracranial Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI changed institutions
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Julius Chapiro, Associate Professor of Radiology, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000031462; 1R21CA259964-01A1 (NIH)
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Cancer Head Neck; Metastatic Cancer; Metastatic Lung Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasm Metastasis; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with head and neck squamous cell carcinoma who plan to undergo tumor resection and lymph node resection (Aim1). Patients with metastases to the brain from melanoma, lung cancer, breast cancer (Aim 2).12 patients with head and neck cancer will be recruited for Aim 1. 12 patients with brain metastases will be recruited for Aim 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Head and neck cancer (Experimental): Participants with head and neck squamous cell carcinoma who plan to undergo tumor resection and lymph node resection.
  Interventions: Drug: adnectin 18F-BMS-986192 Head and Neck Cancer
- Brain Metastases (Experimental): Participants with metastases to the brain from melanoma, lung cancer, breast cancer.
  Interventions: Drug: adnectin 18F-BMS-986192 Brain Metastases

INTERVENTIONS:
Drug: adnectin 18F-BMS-986192 Head and Neck Cancer — Head and Neck Cancer: PET imaging will be performed after initial diagnosis and within 2 weeks of MRI or CT of the neck done as standard of care. MRI will include T1 weighted pre and post gadolinium spin echo, diffusion weighted imaging, and T2 weighted imaging. CT of the head and neck with contrast will be performed per standard clinical protocol. Patients will get one intravenous line and one radial artery line placed prior to imaging and up to 5.5mCi (204MBq) of [18F] PDL192 tracer will be administered intravenously, as a bolus, once the patient is positioned on the scanner. 42 PET data will be acquired at single bed position and in list mode for 120 min after the start of tracer administration. Samples will be drawn from radial artery line.
  Other Names: [18F]PDL192
  Arms: Head and neck cancer
Drug: adnectin 18F-BMS-986192 Brain Metastases — Brain Metastases: Recruited patients will undergo standard clinical MRI within 2 weeks prior to PET, including T1 weighted pre- and post-gadolinium spin-echo and gradient-echo imaging, diffusion weighted imaging, susceptibility weighted imaging (2D SWI), T2 weighted imaging, 3D FLAIR, and combined DCE and dynamic susceptibility contrast (DSC) perfusion (DCE perfusion will be performed first, DSC perfusion will utilize T2 spin echo images). DCE perfusion will be processed on syngo Tissue 4D software (Siemens). DSC perfusion will be processed with syngo MR Perfusion Engine (Siemens). Patients will get one intravenous line and one radial artery line placed prior to imaging and up to 5.5mCi (204MBq) of [18F] PDL192 tracer will be administered intravenously, as a bolus, once the patient is positioned on the scanner. 42 PET data will be acquired at single bed position and in list mode for 120 min after the start of tracer administration. Samples will be drawn from radial artery line.
  Other Names: [18F]PDL192
  Arms: Brain Metastases

SUMMARY:
This study aims to determine the feasibility of non-invasive quantitative PD-L1 measurement using [a novel PD-L1 positron emission tomography (PET) tracer and perform immunohistochemistry based measurement of PD-L1 levels within resected lesions in head and neck cancer and brain metastases.

DETAILED DESCRIPTION:
This study aims to validate a non-invasive quantitative imaging method of whole tumors using a novel PD-L1 positron emission tomography (PET) tracer in patients with head and neck cancer who undergo resection of primary tumor and locoregional lymph node metastases thus providing an excellent model to perform correlative studies with immunohistochemistry (IHC).

The investigators will extend the study to patients with brain metastases because there is a critical need for a non-invasive test for PD-L1 in this population, as biopsy of these lesions is rare.

In this study, the investigators will image patients with brain metastases, which are predominantly from lung cancer and melanoma, that are planned to undergo biopsy. The ultimate goal of this research is to validate quantitative PD-L1 PET imaging in determining PD-L1 expression within primary and metastatic cancer without the need for biopsy and identify parameters of PD-L1 quantitative PET that will allow its translation into clinical practice. This method can then be used to determine which patients may benefit from immunotherapy.

The primary objective of this study aims to test the difference in non-invasive quantitative PD-L1 PET measures (VT) of lesions between different groups of PD-L1 levels (PD-L1 ≥90% vs <1%) in head and neck cancer primary lesions.

Secondary objectives:

1. To establish lesion level association between immunohistochemistry measures of PD-L1 levels within primary head and neck cancer lesions (as the outcome) and PD-L1 PET measures (VT);
2. To establish lesion level association between immunohistochemistry measures of PD-L1 levels within locoregional metastases within the neck and resected normal lymph nodes (as the outcome) and PD-L1 PET measures (VT).
3. To establish lesion level association between the degree of tumor inflammatory cell infiltration on IHC in primary head and neck squamous cell carcinoma (SCC) lesions (as the outcome) and PD-L1 PET measures (VT);
4. To establish lesion level association between the degree of tumor inflammatory cell infiltration on IHC in metastatic head and neck SCC lesion (as the outcomes) and PD-L1 PET measures (VT).

Tertiary objective:

To establish lesion level correlation of IHC measures of total/tumor/inflammatory cell PD-L1 levels to PD-L1 (VT) on PET in brain metastases

ELIGIBILITY:
Inclusion Criteria for Head and Neck Cancer:

* Patients with resectable squamous cell carcinoma of the oropharynx (HPV positive and HPV negative).
* Resectability will be confirmed by a surgical co-investigator.
* If available, HPV-association determined by institutional p16 testing (CINtec antibody demonstrating strong and diffuse nuclear and cytoplasmic staining is at least 70% of cells).
* Absolute neutrophil count (ANC) > 1500/microliter, absolute lymphocyte count (ALC) >1000/microliter, hemoglobin > 9 g/dl, platelets > 100,000/microliter.
* aspartate aminotransferase (AST) and alanine transaminase (ALT) < 5 x upper limit of normal. Bilirubin < 1.5 x upper limit of normal.
* Albumin > 0 g/dl.
* Creatinine < 5 x upper limit of normal.
* Women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to treatment

Inclusion Criteria for Brain Metastases:

* Patients with brain metastases
* Tumor size equal or greater than 1 cm
* Resectability or need for laser interstitial thermal therapy (LITT) will be confirmed by a surgical co-investigator.
* Absolute neutrophil count (ANC) > 1500/microliter, absolute lymphocyte count (ALC) >1000/microliter, hemoglobin > 9 g/dl, platelets > 100,000/microliter
* AST and ALT < 5 x upper limit of normal. Bilirubin < 1.5 x upper limit of normal.
* Albumin > 0 g/dl.
* Creatinine < 5 x upper limit of normal.
* Women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to treatment

Exclusion Criteria for Head and Neck Cancer:

* Medical contraindication to surgery.
* Full dose anticoagulation.
* Concomitant invasive malignancy, or malignancy within 2 years except for hormonally responsive breast or prostate cancer, resected non-melanoma skin cancer, resected uterine cervical carcinoma.
* Inability to give informed consent.
* Prior systemic therapy, radiation or gross resection for the tumor under study.
* Women may not be pregnant or breast-feeding.
* Receipt of other systemic therapy including investigational agents, radiation or gross resection for treatment of the tumor under study.

Exclusion Criteria for Brain Metastases:

* Medical contraindication to brain surgery.
* Full dose anticoagulation.
* Inability to give informed consent.
* Women may not be pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Non-invasive quantitative PD-L1 levels will be measured using PET measures (VT) of lesions for the groups of PD-L1 levels (PD-L1 ≥90% vs <1%, PD-L1 ≥50% vs <1%) in head and neck cancer primary lesions | from with in 2 weeks perioperative up to postoperative
  To test the difference in non-invasive quantitative PD-L1 PET measures (VT) of lesions between different groups of PD-L1 levels (PD-L1 ≥90% vs <1%) in head and neck cancer primary lesions

SECONDARY OUTCOMES:
Immunohistochemistry vs PET measure of PD-L1 levels in head and neck cancer primary lesion | from with in 2 weeks perioperative up to postoperative
  To establish lesion level association comparing immunohistochemistry measures of PD-L1 levels within primary head and neck cancer lesions and PD-L1 PET measures (VT) using Pearson correlation between pathology based measure and imaging based measure.
Immunohistochemistry vs PET measure of PD-L1 levels in head and neck cancer locoregional neck metastatic lesions and resected normal lymph nodes | from with in 2 weeks perioperative up to postoperative
  To establish lesion level association comparing immunohistochemistry measures of PD-L1 levels within locoregional metastases within the neck and resected normal lymph nodes (as the outcome) and PD-L1 PET measures (VT) using Pearson correlation between pathology based measure and imaging based measure.
Immunohistochemistry vs PET measure of infiltrating inflammatory cells in head and neck cancer primary lesion | from with in 2 weeks perioperative up to postoperative
  To establish lesion level association comparing the degree of tumor inflammatory cell infiltration seen on IHC in primary head and neck SCC lesions (as the outcome) and PD-L1 PET measures (VT) using Pearson correlation between pathology based measure and imaging based measure.
Immunohistochemistry vs PET measure of infiltrating inflammatory cells in head and neck cancer locoregional neck metastatic lesions and resected normal lymph nodes | from with in 2 weeks perioperative up to postoperative
  To establish lesion level association comparing the degree of tumor inflammatory cell infiltration on IHC in metastatic head and neck SCC lesion (as the outcomes) and PD-L1 PET measures (VT) using Pearson correlation between pathology based measure and imaging based measure.

OTHER OUTCOMES:
Immunohistochemistry vs PET measure of PD-L1 levels within resected brain metastasis tumor cells | from with in 2 weeks perioperative up to postoperative
  To establish lesion level correlation of IHC measures of total/tumor/inflammatory cell PD-L1 levels compared to PD-L1 (VT) on PET in brain metastases using Pearson correlation between pathology based measure and imaging based measure.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam S Aboian, MD PhD, Principal Investigator — Yale University
Locations (1):
- Yale University PET Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No